CLINICAL TRIAL: NCT00763061
Title: A Twelve-Week, Double Masked, Parallel Group, Study of Travoprost 0.004% Compared to Timolol 0.5% in Patients With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Travatan Versus Timoptic in Treating Open-angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Benny Li, Ph.D., Alcon Research Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-06-02
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2010-01-26 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Travoprost; Ophthalmic Solutions; Timolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Travoprost 0.004% (Experimental): Travoprost 0.004%
  Interventions: Drug: Travoprost 0.004% Ophthalmic Solution (Travatan)
- Timolol 0.5% (Active Comparator): Timolol 0.5%
  Interventions: Drug: Timolol 0.5% Ophthalmic Solution (Timoptic)

INTERVENTIONS:
Drug: Travoprost 0.004% Ophthalmic Solution (Travatan) — Travoprost at 9 AM + Placebo & 9 PM
  Arms: Travoprost 0.004%
Drug: Timolol 0.5% Ophthalmic Solution (Timoptic) — Timolol in each eye, twice daily at 9 AM & 9 PM
  Arms: Timolol 0.5%

SUMMARY:
To evaluate the Intraocular Pressure (IOP) lowering efficacy and safety of Travoprost 0.004% compared to Timolol 0.5% in patients with open-angle glaucoma (OAG) or ocular hypertension (OH). The study structure is a parallel design. The patients will receive treatment for 12 weeks.

DETAILED DESCRIPTION:
To evaluate the IOP lowering efficacy and safety fo Travoprost 0.004% compared to Timolol 0.5% in patients with open-angle glaucoma (OAG) or ocular hypertension (OH). The study structure is a parallel design. The patients will receive treatment for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years;
* IOP=16-30mmHg
* OH or OAG with visual filed abnormality:

  1. ≥3 adjacent points in 24 degrees field on the same side of the horizontal meridian, that have p <5% on the prepapillary diameter plot, one of which must have p <1%,
  2. Glaucoma Hemifield Test outside normal limits,
  3. Corrected Pattern Standard Deviation with p <5%

Exclusion Criteria:

* Previous damage of anterior chamber angle;
* ocular inflammation or ocular surgery within the past 3 months; Best Corrected Visual Acuity (logMAR) <1.0;
* contact lens wearer;
* severe central field loss;
* uncontrolled cardiovascular, hepatic or renal disease;
* any medication within past 1 month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2006-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 111 patients were enrolled in this study at 4 hospitals
Pre-assignment Details: Eligibility patients were washed out for up to 4 weeks before randomization
Groups:
- Travoprost 0.004%: Travoprost at 9 AM + Placebo & 9 PM
- Timolol 0.5%: Timolol in each eye, twice daily at 9 AM & 9 PM
Period: Overall Study
Arm/Group | Travoprost 0.004% | Timolol 0.5%
Started | 54 | 57
Completed | 49 | 44
Not Completed | 5 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Travoprost 0.004% | Timolol 0.5% | Total
Number analyzed (Participants) | 54 | 57 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 33 | 31 | 64
  >=65 years | 19 | 25 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 26 | 48
  Male | 32 | 31 | 63

OUTCOME MEASURES:

1. Primary Outcome: Mean Intraocular Pressure (IOP) at 9 AM
Description: Bilateral IOP measurements by Goldmann applanation were performed at 9AM and 4 PM. Two IOP measurements were taken and averaged. If the difference between the first and second reading was greater than 4 mmHg, a third reading was taken and the two nearest readings averaged.
Time Frame: At Week 12 - At the 9 AM time point for the patient's worse eye.
Measure: Mean (Standard Deviation); unit: millimeters mercury (mmHg)
Arm/Group | Travoprost 0.004% | Timolol 0.5%
Number analyzed (Participants) | 49 | 44
millimeters mercury (mmHg) | 16.3 (4.27) | 18.1 (4.32)

2. Secondary Outcome: Mean IOP Change From Baseline at 9 AM
Description: as for outcome 1
Time Frame: Baseline to Week 12 - at 9 AM
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Travoprost 0.004% | Timolol 0.5%
Number analyzed (Participants) | 49 | 44
mmHg | -5.1 (4.35) | -4.4 (4.35)

3. Primary Outcome: Week 12 - Mean IOP At 4 PM
Description: as for outcome 1
Time Frame: At the 4 PM time point for the patient's worse eye.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Travoprost 0.004% | Timolol 0.5%
Number analyzed (Participants) | 49 | 44
mmHg | 15.7 (3.16) | 17.9 (4.02)

4. Secondary Outcome: Mean IOP Change at 4 PM
Description: as for outcome 1
Time Frame: Baseline to Week 12 - at 4 PM
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Travoprost 0.004% | Timolol 0.5%
Number analyzed (Participants) | 49 | 44
mmHg | -5.3 (3.69) | -3.7 (4.15)

ADVERSE EVENTS:
Arm/Group | Travoprost 0.004% | Timolol 0.5%
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/57
Other Adverse Events (participants affected / at risk) | 0/54 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No